CLINICAL TRIAL: NCT03862781
Title: Randomized Trial of Intra-Corporeal Anastomosis for RighT Colectomies (RICART Study)
Brief Title: Intra-Corporeal Anastomosis Result in Quicker Return of Bowel Function/Earlier Discharge
Acronym: RICART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Corewell Health West (Other)
Responsible Party: Principal Investigator, James W. Ogilvie, Colorectal Surgeon, Corewell Health West
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2018-139
Record Dates: First submitted 2019-02-05; First posted 2019-03-05 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Disorders

STUDY DESIGN:
Intervention Model Description: After the participants have been consented to the study, the study coordinator will refer to the randomization schedule, and alert the surgeon whether creation of the anastomosis will be done in either an intra-corporeal or extra-corporeal fashion.
Who Masked: Participant
Masking Description: The patients, nursing staff and the perioperative care team (physician assistants, residents) will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intra-corporeal (Other): Right Hemicolectomy
  Interventions: Procedure: Right Hemicolectomy
- Extra-corporeal (Other): Right Hemicolectomy
  Interventions: Procedure: Right Hemicolectomy

INTERVENTIONS:
Procedure: Right Hemicolectomy — Minimally invasive approach (robotic or laparoscopic) with the creation of an anastomosis.

SUMMARY:
Adult patients who are regularly scheduled to undergo a right hemicolectomy via a minimally invasive approach (robotic or laparoscopic) with the creation of an anastomosis.

DETAILED DESCRIPTION:
The purpose of this trial is to investigate whether minimally invasive right colectomies done with an intra-corporeal anastomosis result in quicker return of bowel function and earlier discharge. The primary endpoint of this study will be return of bowel function as measured by passage of flatus and bowel motions. The secondary endpoints will be inpatient length of stay, incision length, postoperative narcotic use, surgical site infection (superficial, deep and organ-space), perioperative morbidity and operating room charges.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients are those over 18 years of age who are regularly scheduled to undergo a right hemicolectomy via a minimally invasive approach (robotic or laparoscopic) with the creation of an anastomosis. Right colectomy will be defined as removal of the ascending colon, ligation of the ileocolic artery and vein, +/- removal of the terminal ileum, +/- removal of the proximal transverse colon, and +/- removal of the right branch of the middle colic artery and vein.

Exclusion Criteria:

* Pregnant women
* Additional colon resection is planned (i.e. left colectomy or proctectomy)
* Vulnerable populations such as prisoners or adults unable to give consent
* If the scheduled surgery is planned at Butterworth hospital (as to standardize the nursing care received postoperatively)
* Emergent cases

Patients will be excluded from the study intra-operatively if:

* The procedure is converted to an open resection
* If a loop ileostomy is performed in addition to the right colectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2019-01-28 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Return of bowel function | up to 2 weeks
  Flatus and bowel motions

SECONDARY OUTCOMES:
Inpatient length of stay | up to 2 weeks
  Days in the hospital after surgery
Incision length | Surgery date
  cm's
Postoperative narcotic use | up to 2 weeks
  Average pain scores over first 5 hospital days
Surgical site infection | up to 6 weeks
  (superficial, deep and organ-space)
Perioperative morbidity | Baseline (Prior to surgery)
  Disease state
Operating room charges | Surgery date
  Fees for operating room

CONTACTS AND LOCATIONS:
Overall Officials: James W Ogilvie, Jr., MS, Principal Investigator — Corewell Health West
Locations (1):
- Spectrum Health Medical Group, Grand Rapids, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to Share IPD.

DOCUMENTS (1):
  • Informed Consent Form (2025-05-20): https://cdn.clinicaltrials.gov/large-docs/81/NCT03862781/ICF_005.pdf